CLINICAL TRIAL: NCT05820542
Title: Comparison of Glottic Opening Percentage (POGO) With Miller and McGrath MAC Videoingoscopes According to Direct Epiglottis Lifting Method
Brief Title: Glottic Opening Percentage (POGO) With Miller and McGrath MAC Videoingoscopes
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2022/14
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Endotracheal intübation
Keywords: percentage of glottic opening; laryngoscopy; direct epiglottis lifting method

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group M (n=42), Miller laryngoscope: The effect of direct epiglottis lifting method on the percentage of glottic patency in Miller and McGraht laryngoscopy.
  Interventions: Other: miller laryngoscope
- Group V (n= 43), McGrath MAC videolaryngoscope: The effect of direct epiglottis lifting method on the percentage of glottic patency in Miller and McGraht laryngoscopy.
  Interventions: Other: McGrath MAC videolaryngoscope

INTERVENTIONS:
Other: miller laryngoscope — The percentage of glottic opening (POGO) will be evaluated according to the method of lifting the epiglottis (direct imaging).
  Groups: Group M (n=42), Miller laryngoscope
Other: McGrath MAC videolaryngoscope — The percentage of glottic opening (POGO) will be evaluated according to the method of lifting the epiglottis (direct imaging).
  Groups: Group V (n= 43), McGrath MAC videolaryngoscope

SUMMARY:
The aim of this study is to compare the percentage of glottic opening (POGO) with Miller and McGrath MAC Videoingoscopes compared to the direct epiglottis lifting method.

DETAILED DESCRIPTION:
The aim of this study is to compare the percentage of glottic opening (POGO) with Miller and McGrath MAC Videoingoscopes compared to the direct epiglottis lifting method.

ELIGIBILITY:
Inclusion Criteria:

* Those who agreed to participate in the study
* He will undergo elective surgery
* Endotracheal intubation required
* 18-65 years old
* ASA 1-2 risk
* Body mass index<30
* No risk of difficult intubation

Exclusion Criteria:

* Those who do not want to participate in the study,
* Allergic to study drugs,
* Pregnant women
* Those with a history of difficult intubation
* They will be applied rapid-serial intubation
* Emergency

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 85 patients 18-65 years both genders in all surgeries requiring intubation
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Glottic Opening Percentage (POGO) With Miller and McGrath MAC Videolaryngoscopes According to Direct Epiglottis Lifting Method | during laryngoscopy
  Comparison of Glottic Opening Percentage (POGO) With Miller and McGrath MAC Videolaryngoscopes According to Direct Epiglottis Lifting Method

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided